CLINICAL TRIAL: NCT05330767
Title: DermaClose Continuous External Tissue Expander for the Management of Four-Compartment Fasciotomy and Full-Thickness Wounds.
Brief Title: DermaClose DUKE Fasciotomy and Wound Study
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: BXU568622
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Wound of Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Wound on either the upper or lower extremity with DermaClose and/or DermaClose XL: Non-fasciotomy
  Interventions: Device: DermaClose Continuous External Tissue Expander Device; Device: DermaClose XL Continuous External Tissue Expander Device
- Wound undergoing fasciotomy with DermaClose and/or DermaClose XL
  Interventions: Device: DermaClose Continuous External Tissue Expander Device; Device: DermaClose XL Continuous External Tissue Expander Device
- Wound undergoing fasciotomy with conventional wound dressings
  Interventions: Device: Conventional wound dressings

INTERVENTIONS:
Device: DermaClose Continuous External Tissue Expander Device — Constant tension and self-tensioning device. Supplied sterile and for single use only.
  Groups: Wound on either the upper or lower extremity with DermaClose and/or DermaClose XL; Wound undergoing fasciotomy with DermaClose and/or DermaClose XL
Device: DermaClose XL Continuous External Tissue Expander Device — Intended for large wounds that are greater than 8 cm in width. Constant tension and self-tensioning device. Supplied sterile and for single use only
  Groups: Wound on either the upper or lower extremity with DermaClose and/or DermaClose XL; Wound undergoing fasciotomy with DermaClose and/or DermaClose XL
Device: Conventional wound dressings — Wet-to-dry, gauze, and negative pressure wound therapy.
  Groups: Wound undergoing fasciotomy with conventional wound dressings

SUMMARY:
To evaluate the clinical performance of DermaClose and DermaClose XL Continuous External Tissue Expander (CETE) devices to reduce wound size and/or assist with closure in acute full thickness wounds of the skin and assess the need for skin grafting for patients undergoing a four-compartment leg fasciotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age at the time of consent.
* Patient with a full thickness acute wound(s) of the skin:

  1. On either the upper or lower extremity (including four-compartment leg fasciotomy), in whom DermaClose and/or DermaClose XL is applied during surgery, OR
  2. Undergoing a four-compartment leg fasciotomy requiring conventional wound dressing.
* Patient has signed a written informed consent form (ICF) per 21 Code of Federal Regulations (CFR) Part 50.55(e).

Exclusion Criteria:

* Patient in whom the product was used off-label (except for patients who have the device on for longer than 14 days)
* Patient with wound(s) that exhibit any of the following:

  * Ischemic tissue,
  * Infected tissue,
  * Acute burned tissue,
  * Fragile tissue at the edges of the wound(s).
* Patient, who in surgeon's opinion, does not fit the criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who have acute full thickness wound(s) of the skin (including four-compartment leg fasciotomy) and in whom DermaClose and/or DermaClose XL, or conventional dressing is used.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Proportion of investigator-confirmed wound size reduction or assistance with closure of acute full thickness wounds | Up to 14 Days (or longer if deemed necessary by surgeon)
  Wounds may result from four-compartment leg fasciotomies.

SECONDARY OUTCOMES:
Mean percentage of wound size reduction | Up to 14 Days (or longer if deemed necessary by surgeon)
  Calculated at time of device removal.
Median number of days until wound closure | Up to 14 Days (or longer if deemed necessary by surgeon)
  Defined as the ability to complete surgical closure.
Proportion of wounds treated with subsequent reconstruction with a skin graft after fasciotomy | Up to 60 Days
  Plastic surgery may be consulted for reconstruction by the referring surgeon, or the patient may be recommended for study inclusion by the referring surgeon who plans on using conventional dressing to manage the wound(s).
Proportion of wounds requiring subsequent surgical procedure(s) for wound closure | Up to 60 Days
  Includes participants with conventional closure modality or skin graft
Number of days until hospital discharge | Up tp 60 Days
  Median time (min, max) in days will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: https://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy